CLINICAL TRIAL: NCT07320937
Title: Effects of Yiqi Fuyuan Paste Formula in Chronic Fatigue Syndrome: A Randomized Double-Blind Controlled Clinical Trial.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Xiao tian zhang, Director of the Preventive Health Center, ShuGuang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1603-186-01
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: CFS

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo, oral, twice daily for 8 weeks
  Interventions: Other: Placebo(a look-alike substance that contains no drug)
- "Yiqi Fuyuan Paste Formula" test group (Experimental): Yiqi Fuyuan Paste Formula, oral, twice daily for 8 weeks
  Interventions: Other: "Yiqi Fuyuan Paste Formula" test group

INTERVENTIONS:
Other: "Yiqi Fuyuan Paste Formula" test group — The intervention is a custom-made herbal paste prepared from food-medicine homology ingredients, including Astragalus membranaceus, Codonopsis pilosula, Dioscorea opposita, and others. It is administered orally twice daily for 12 weeks to improve immune function and quality of life in patients with chronic fatigue or post-illness recovery.
  Method of taking the ointment: Start taking it from the time it is prepared. It is generally recommended to take it on an empty stomach. The total duration of taking it is 8 weeks (20g per dose, twice a day), taking it warm in the morning and evening respectively; The ointment should be stored in the refrigerator for refrigeration.
  Arms: "Yiqi Fuyuan Paste Formula" test group
Other: Placebo(a look-alike substance that contains no drug) — Method of taking the ointment: Start taking it from the time it is prepared. It is generally recommended to take it on an empty stomach. The total duration of taking it is 8 weeks (20g per dose, twice a day), taking it warm in the morning and evening respectively; The ointment should be stored in the refrigerator for refrigeration.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if "Yiqi Fuyuan Paste Formula" (a traditional Chinese medicinal paste made from medicinal and edible Chinese medicines and health food like Ginseng Radix et Rhizoma, Astragali Radix et Rhizoma, Codonopsis Radix, Atractylodis Macrocephalae Rhizoma, Poria Cocos, Coicis Semen, Dioscoreae Rhizoma, Nelumbinis Semen, Angelicae Sinensis Radix, Lycii Fructus, Citri Reticulatae Pericarpium, Juglandis Semen, Longan Arillus, Sesami Nigri Semen, Jujubae Fructus, Glycyrrhizae Radix et Rhizoma, and fine ingredients) works to ease Chronic Fatigue Syndrome (CFS) symptoms in adults. It will also learn about the safety of "Yiqi Fuyuan Paste Formula". The main questions it aims to answer are:

1. Does "Yiqi Fuyuan Paste Formula" help reduce CFS-related fatigue (measured by the Fatigue Assessment Instrument, FAI)
2. What underlying bodily changes (shown in blood tests) might explain its effects.

Researchers will compare "Yiqi Fuyuan Paste Formula" to a placebo (a look-alike substance that contains no drug) to see if "Yiqi Fuyuan Paste Formula" works to ease CFS symptoms.

Participants will:

1. Take "Yiqi Fuyuan Paste Formula" or a placebo every day for 2 months
2. Visit the clinic before and after the intervention for checkups and tests
3. Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 - 65 years old, gender not restricted;

  * Patients meeting the diagnostic criteria for chronic fatigue syndrome;

    * Patients identified as having an "qi deficiency" or "balanced" constitution according to traditional Chinese medicine body type assessment; ④ Voluntary participants who have signed the informed consent form.

Exclusion Criteria:

Those who have any of the following conditions will not be included in this trial.

* Those with severe depression or other mental disorders, as well as severe diseases of the heart, brain, liver, kidney and hematopoietic system; ② Those who are known to be allergic to the ingredients used in the ointment and have a severe allergic constitution;

  * Women who are currently breastfeeding, pregnant or have the intention to get pregnant during the trial period; ④ Those who are currently participating in other medical clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
FAI (Fatigue Assessment Instrument) | week4

SECONDARY OUTCOMES:
SF-36 (The MOS 36-Item Short-Form Health Survey) | week4
QDC（Qi deficiency constitution score） | week4

OTHER OUTCOMES:
inflammatory factors | week 4
  Changes in inflammatory factors(IL-2, IL-6, IL-10, IgA, IgM, INF-γ TNF-α) through peripheral serum
Differential genes | week 4
  Screening of differentially expressed genes through RNA-seq

CONTACTS AND LOCATIONS:
Locations (1):
- Shuguang hospital, Shanghai, Pudong New Area, China

IPD SHARING:
Plan to Share IPD: No